CLINICAL TRIAL: NCT04555837
Title: A Phase I-II, Open Label Study Evaluating the Safety and Efficacy of Alisertib and Pembrolizumab in Patients With Rb-Deficient Head and Neck Squamous Cell Carcinomas
Brief Title: Alisertib and Pembrolizumab for the Treatment of Patients With Rb-deficient Head and Neck Squamous Cell Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0210; NCI-2020-05051 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0210 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Malignant Solid Neoplasm
Keywords: head and neck cancer; HPV; Immunotherapy; squamous cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — MLN 8237; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (alisertib, pembrolizumab) (Experimental): Patients receive alisertib PO BID on days 1-7 and pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alisertib; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Alisertib — Given PO
  Other Names: Aurora A Kinase Inhibitor MLN8237; MLN-8237; MLN8237
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase I/II trial investigates the best dose and effect of alisertib in combination with pembrolizumab in treating patients with Rb-deficient head and neck squamous cell cancer. Alisertib may help block the growth of cancer.. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the tumor, and may interfere with the ability of tumor cells to grow and spread. Giving alisertib in combination with pembrolizumab may help control Rb-deficient head and neck squamous cell cancer. HPV positive head and neck cancers are Rb-deficient.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommend phase II dose of the combination of alisertib and pembrolizumab. (Phase I) II. To determine the overall response rate (ORR) and progression free survival (PFS) of patients with recurrent or metastatic Rb-deficient head and neck squamous cell carcinoma (HNSCC) treated with the combination of pembrolizumab and alisertib. (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate the safety of the combination of pembrolizumab and alisertib in patients with solid tumors.

II. To determine the overall survival in HNSCC patients treated with the combination of pembrolizumab and alisertib.

III. To determine the relationship between pharmacokinetics, pharmacodynamics, baseline immune and tumor biomarkers and clinical responses in patients treated with alisertib and pembrolizumab.

IV. To determine correlations between clinical responses and the effect of the treatment on human papilloma virus (HPV)-reactive T cells in HPV+ cancers.

V. To determine correlations between clinical responses and tumor infiltrating lymphocyte function and T cell repertoire.

OUTLINE: This is a phase I, dose-escalation study of alisertib in combination with fixed dose pembrolizumab followed by a phase II study.

Patients receive alisertib orally (PO) twice daily (BID) on days 1-7 and pembrolizumab intravenously (IV) over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2-3 months.

ELIGIBILITY:
Inclusion Criteria - phase II only

1. Histologically or cytological confirmed diagnosis of Rb-deficient HNSCC for which no standard curative therapy is available.
2. Rb deficient HNSCC includes CLIA-certified testing confirming one of the following:

A. HPV positive as determined by any one of the following: p16 immunohistochemistry (IHC), HPV RNA in situ hybridization (ISH), RNAscope (mRNA ISH), DNA ISH, DNA PCR, or qRT PCR.

B. No Rb protein expression in the tumor as determined by IHC.41, 48 3. Progression on prior treatment with an anti-PD-1 antibody or an anti-PD-L1 antibody.

A. Has received at least 2 doses of a PD-1/PD-L1 checkpoint blockade therapy. B. Clinical or radiographical progression has been documented within 12 weeks from the last dose of PD-1/PD-L1 checkpoint blockade therapy.

Inclusion Criteria - phase I only

1. Histologically or cytological confirmed diagnosis of an invasive solid tumor malignancy, for which no standard curative or life prolonging therapy is available.

Inclusion Criteria - both phase I and phase II

1. Male or female patients ≥ 18 years of age.
2. ECOG performance status of ≤ 2 (see section 7.4).
3. Clinical laboratory values as specified below within 22 days before the first dose of study drug

   * Absolute neutrophil count (ANC) > 1500/mm³
   * Platelets > 100,000/mm³
   * Hgb > 9 g/dL. Values must be obtained without need for myeloid growth factor or platelet transfusion support within 14 days, however, erythrocyte growth factor is allowed as per published ASCO guidelines.
   * Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
   * SGOT (AST) and SGPT (ALT)< 2.5 x ULN. AST and/or ALT may be up to 5X ULN if with known liver mets or total 3 x ULN with direct bilirubin ≤ ULN in patients with well-documented Gilbert syndrome.
   * Adequate renal function as defined by calculated creatinine clearance ≥30 ml/min (Cockroft-Gault Formula, see Section 7.5).
4. Measurable disease according to RECIST version 1.1.
5. Voluntary written consent must be given before performance of any study related procedure not part of standard of care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
6. Patients must be able to either swallow alisertib enteric coated tablets, swallow alisertib oral solution formulation, or administer alisertib oral solution formulation via a feeding tube that terminates in the stomach.
7. Willing to provide blood and tissue for correlative research purposes.
8. Female patients who:

   * Are postmenopausal for at least 1 year before the screening visit, OR
   * Are surgically sterile, OR
   * If they are of childbearing potential, agree to practice 1 highly effective method of contraception and 1 additional effective (barrier) method at the same time, from the time of signing the informed consent through 120 days after the last dose of study drug, OR
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)
9. Male patients, even if surgically sterilized (i.e., status postvasectomy), who:

   * Agree to practice effective barrier contraception during the entire study treatment period and through 120 after the last dose of study drug, OR
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)

Exclusion Criteria:

1. Radiation therapy to more than 25% of the bone marrow. Whole pelvic radiation is considered to be over 25%.
2. Prior allogeneic bone marrow or organ transplantation.
3. Known gastrointestinal (GI) disease or GI procedures that could interfere with the oral absorption or tolerance of alisertib. Examples include, but are not limited to partial gastrectomy, history of small intestine surgery, and celiac disease.
4. Inability to swallow (or use a feeding tube to administer) oral medication or inability or unwillingness to comply with the administration requirements related to alisertib.
5. Known history of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness, such as severe chronic obstructive pulmonary disease; requirement for supplemental oxygen.
6. Requirement for constant administration of proton pump inhibitor, H2 antagonist, or pancreatic enzymes throughout the study. The intermittent use of H2-antagonists and antacids (including carafate) is only allowed within these guidelines:

   1. H2 antagonists until D-1 and after the dosing of alisertib is done
   2. Antacid formulations until 2 hours before doing and after 2 hours following dosing.
   3. PPI is allowed until D-5 of first alisertib dose. PPIs are prohibited throughout the study
7. Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see Section 7.3), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
8. Female subject who is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative urine or serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
9. Female patient who intend to donate eggs (ova) during the course of this study or 120 days after receiving their last dose of study drug(s).
10. Male patients who intend to donate sperm during the course of this study or 120 days after receiving their last dose of study drug(s).
11. Other severe acute or chronic medical or psychiatric condition, including uncontrolled diabetes, malabsorption, resection of the pancreas or upper small bowel, requirement for pancreatic enzymes, any condition that would modify small bowel absorption of oral medications, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for enrollment in this study.
12. Diagnosed or treated for another invasive malignancy within 2 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
13. Has received any anti-cancer treatment including investigational agents within 21 days prior to first dose of alisertib.
14. Patients who receive gamma knife radiosurgery for brain metastases or whole brain radiation are eligible if gamma knife radiosurgery was completed > 2 weeks before treatment is started or whole brain radiation was performed > 4 weeks before treatment is started, and are clinically stable (not requiring steroids or anti-epileptic drugs).
15. Known hypersensitivity to any of the excipients of alisertib enteric coated tablets or severe reaction to any human monoclonal antibody.
16. Patients with a prior history of clinically significant metabolic acidosis (exclusion only for patients receiving alisertib oral solution).
17. Major surgery within 28 days prior to first dose of alisertib or persisting side effects that have not improved to NCI-CTCAE grade 1 or better.
18. Patients who are on (or will require) prolonged systemic corticosteroid treatment during the study except for replacement dosing for adrenal insufficiency.
19. Concurrent severe and/or uncontrolled medical conditions that would, in the investigator's judgment, contraindicate patient participation in the clinical study or require concomitant anti-cancer drugs (e.g. active or uncontrolled severe infection, chronic active hepatitis, immuno-compromised, acute or chronic pancreatitis, uncontrolled high blood pressure, interstitial lung disease).
20. Patients with active, known, diagnosed or suspected autoimmune disease. Patients suffering from vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring thyroid hormone replacement therapy, or psoriasis not requiring systemic treatment can be enrolled.
21. Patients diagnosed with active interstitial lung disease (ILD)/pneumonitis or a history of ILD/pneumonitis or another condition requiring immunosuppressive doses of systemic medication such as systemic corticosteroids or absorbed topical corticosteroids (doses ≥ 10 mg/day prednisone or equivalent) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical corticosteroids, adrenal replacement doses, or < 10 mg daily prednisone or equivalent are permitted.
22. Administration of any live vaccine within 30 days before first dose of study drug.
23. Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B virus or hepatitis C virus, except for: Patients with HIV who have controlled infection (undetectable viral load and CD4 count above 350 cells/mm3 either spontaneously or on a stable antiviral regimen) are permitted; Patients with hepatitis B (HepBsAg+) virus who have controlled infection (serum hepatitis B virus DNA PCR that is below the limit of detection AND receiving antiviral therapy for hepatitis B) are permitted; Patients who are hepatitis C virus antibody positive (HCV Ab +) who have controlled infection (undetectable HCV RNA by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy) are permitted.
24. Participating in another therapeutic clinical trial.
25. Prior immune-related adverse events (irAE) as follows:

A. Any life-threatening irAE will not be eligible.

B. Any grade irAE of the following types will not be eligible:

* i. Nervous system irAE
* ii. Ocular irAE
* iii. Cardiovascular irAE
* iv. Severe Cutaneous Adverse Reactions (SCAR)
* v. Hematological irAE

C. Any grade endocrine irAE will be eligible if replacement therapy can compensate for the resulting deficit.

D. Grade ≥ 2 irAE of the following will not be eligible:

* i. Colitis
* ii. Hepatitis
* iii. Bullous Dermatoses
* iv. Pneumonitis
* v. Musculoskeletal
* vi. Renal

E. Grade ≥ 3 cutaneous irAE will not be eligible.

F. All irAEs must have resolved to Grade ≤ 1 at least 14 days before the planned first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faye M Johnson, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient with Rb-deficient head and neck squamous cell carcinomas. 28 patient were screened for the study. 4 patients were screen failed.
Groups:
- Phase I; Phase II: Pembrolizumab 200mg IV every 3 weeks + Alisertib 40mg PO BID x 7 days every 21 days
Period: Overall Study
Arm/Group | Phase I | Phase II
Started | 10 | 14
Completed | 10 | 12
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II | Total
Number analyzed (Participants) | 10 | 14 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 3 | 7 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 6 | 14 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 14 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 7 | 13 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Phase I: The Recommended Phase II Dose Determenation. Phase II: Overall Response Rate (ORR) and Progression Free Survival (PFS)
Description: Phase I: To determine the recommend phase II dose of the combination of alisertib and pembrolizumab
Time Frame: Approximately 33 months
Population: Phase I: To determine the recommend phase II dose of the combination of alisertib and pembrolizumab
Measure: Number; unit: mg
Arm/Group | Phase I
Number analyzed (Participants) | 10
mg | 40

2. Primary Outcome: Phase II: Overall Response Rate (ORR)
Description: Phase II: To determine the overall response rate (ORR) of patients with recurrent or metastatic Rb-deficient head and neck squamous cell carcinoma (HNSCC) treated with the combination of pembrolizumab and alisertib.
Time Frame: Approximately 33 months
Population: Insufficient number of participants with events
Measure: Count of Participants; unit: Participants
Groups:
- Phase II: Pembrolizumab 200mg IV every 3 weeks + Alisertib 50mg po BID x 7 days every 21 days
Arm/Group | Phase II
Number analyzed (Participants) | 14
Participants | 0

3. Primary Outcome: Phase II: Progression Free Survival (PFS)
Description: Phase II: To determine the progression free survival (PFS) of patients with recurrent or metastatic Rb-deficient head and neck squamous cell carcinoma (HNSCC) treated with the combination of pembrolizumab and alisertib.
Time Frame: Approximately 33 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 14
months | 1.4 [NA to NA] — Insufficient number of participants with events

4. Secondary Outcome: The Safety of the Combination of Pembrolizumab and Alisertib
Description: To evaluate the safety of the combination of pembrolizumab and alisertib in patients with solid tumors.
Time Frame: Adverse events were monitored until off study due to disease progression, death, unacceptable toxicity, consent withdrawal, or physician's discretion, approximately 33 months.
Population: 28 patients (4 patients were screen failures) enrolled from September 2020 to June 2023, 24 were treated and evaluable for safety.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 10 | 14
Participants
  AE | 10 | 13
  SAE | 2 | 2
  Death | 2 | 0

5. Secondary Outcome: The Overall Survival in HNSCC Patients
Description: To determine the overall survival in HNSCC patients treated with the combination of pembrolizumab and alisertib in Phase II only.
Time Frame: 28 patients (4 patients were screen failures) enrolled from September 2020 to June 2023, 24 were treated and evaluable for response. Patients were followed for overall survial for approximately 33 months
Population: To determine the overall survival in HNSCC patients treated with the combination of pembrolizumab and alisertib in Phase II only.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 0 | 14
Months |  | 16.8 [NA to NA] — Insufficient number of participants with events

6. Secondary Outcome: The Relationship Between Pharmacokinetics, Pharmacodynamics, Baseline Immune and Tumor Biomarkers and Clinical Responses
Description: To determine the relationship between pharmacokinetics, pharmacodynamics, baseline immune and tumor biomarkers and clinical responses in patients treated with alisertib and pembrolizumab in phase II only.
Time Frame: The trial design dictated that if there were no objective responses in thefirst cohort of the phase II study, the trial would close after the first cohort.
Population: Data are not collected
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Correlations Between Clinical Responses and the Effect of the Treatment on Human Papilloma Virus (HPV)-Reactive T Cells in HPV+ Cancers.
Description: To determine correlations between clinical responses and the effect of the treatment on human papilloma virus (HPV)-reactive T cells in HPV+ cancers in phase II only.
Time Frame: The trial design dictated that if there were no objective responses in the first cohort of the phase II study, the trial would close after the first cohort.
Population: The trial design dictated that if there were no objective responses in the first cohort of the phase II study, the trial would close after the first cohort. Biopsies were not performed in the first cohort, per study design, and HPV-reactive T cells could not be measured.
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Correlations Between Clinical Responses and Tumor Infiltrating Lymphocyte Function and T Cell Repertoire.
Description: To determine correlations between clinical responses and tumor infiltrating lymphocyte function and T cell repertoire in phase II only.
Time Frame: as for outcome 7
Population: The trial design dictated that if there were no objective responses in the first cohort of the phase II study, the trial would close after the first cohort. Biopsies were not performed in the first cohort, per study design, and tumor infiltrating lymphocyte function and T cell repertoire could not be measured.
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 patients enrolled from September 2020 to June 2023 (4 patients were screen failures), 24 were treated and evaluable for safety. Adverse events were monitored until off study due to disease progression, death, unacceptable toxicity, consent withdrawal, or physician's discretion, approximately 33 months.
Description: All eligible patients who received at least one cycle of treatment were considered evaluable for safety analyses. AEs (realted and unrelated) were graded according to Common Terminology Criteria for AEs version 5.0.
Arm/Group | Phase I | Phase II
All-Cause Mortality (participants affected / at risk) | 2/10 | 0/14
Serious Adverse Events (participants affected / at risk) | 2/10 | 2/14
Other Adverse Events (participants affected / at risk) | 10/10 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (N=10) | Phase II (N=14)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (N=10) | Phase II (N=14)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (11) | 2 (2)
Alkaline phosphatase increased (Investigations) | 3 (10) | 3 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (6) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 9 (35) | 10 (22)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (9) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (3) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 4 (4)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (4) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Creatinine increased (Investigations) | 2 (2) | 3 (4)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Depression (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (8) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry skin (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eye disorders - Other, specify (redness) (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, specify (L upper eye field defects) (Eye disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 9 (13) | 5 (7)
Febrile neutropenia (General disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 1 (1) | 2 (2)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal disorders - Other, specify (complication of Gastric Tube. Replaced at ACCC) (Gastrointestinal disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (Stomach ache) (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (facial cellulitis) (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (Oral Thrush) (General disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (15) | 8 (9)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Hypernatremia (Metabolism and nutrition disorders) | 1 (4) | 1 (1)
Hyperphosphatemia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (6) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (8) | 2 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (4) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 5 (9) | 6 (10)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (4) | 2 (2)
INR increased (Investigations) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1) | 0 (0)
Investigations - Other, specify (Right Shoulder Discomfort) (Investigations) | 1 (1) | 0 (0)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 8 (34) | 10 (28)
Metabolism and nutrition disorders - Other, specify (Vitamin D Deficiency) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Mucositis Oral (Gastrointestinal disorders) | 3 (6) | 4 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 6 (21) | 4 (5)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (3) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (8) | 2 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (skin peeling) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Serpentine rash to bilateral forearms) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Watering eyes (Eye disorders) | 1 (1) | 0 (0)
Weight loss (Investigations) | 3 (4) | 3 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
White blood cell decreased (Investigations) | 7 (35) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT04555837/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-09): https://cdn.clinicaltrials.gov/large-docs/37/NCT04555837/ICF_002.pdf